CLINICAL TRIAL: NCT02806700
Title: Twitter and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01: HL122457-0IA1; R01HL122457-01A1 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Diabetes; Cardiovascular Disease
Keywords: Diabetes; Social Media
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twitter Diabetes Control (No Intervention): This group will be identified as having diabetes from Twitter. This group will be contacted and asked to complete brief surveys
- Twitter Diabetes Intervention (Experimental): This group will be identified as having diabetes from Twitter. This group will be contacted and asked to complete brief surveys. This group will be asked to use twitter for heart health ( e.g. tweeting, following, receiving tweets)
  Interventions: Behavioral: Twitter Diabetes Intervention

INTERVENTIONS:
Behavioral: Twitter Diabetes Intervention — This group will be asked to use twitter for heart health ( e.g. tweeting, following, receiving tweets)
  Arms: Twitter Diabetes Intervention

SUMMARY:
Twitter use is surprisingly well represented across broad demographic population segments and health-related messages. The promise of using Twitter is that its use is growing rapidly, it allows the investigators to view communications that were impossible to intercept before, and it potentially provides information faster and less expensively than collection from other media channels. Prior work also supports that social media interventions can improve health behavior change (e.g. weight loss, physical activity) and outcomes.The overarching goals of this proposal are to understand the uses and limitations of this communication channel to improve patients' ability to manage their CV health condition.

DETAILED DESCRIPTION:
Use Twitter to deliver high impact CV health related content to improve patient activation and disease management for diabetes.

ELIGIBILITY:
Inclusion Criteria:

* diabetes
* uses social media

Exclusion Criteria:

* <21 years of age
* pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Twitter Diabetes Control | Twitter Diabetes Intervention
Started | 316 | 312
Completed | 226 | 252
Not Completed | 90 | 60

BASELINE CHARACTERISTICS:
Population: Total number of participants who completed baseline survey and were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Twitter Diabetes Control | Twitter Diabetes Intervention | Total
Number analyzed (Participants) | 316 | 295 | 611
Age, Continuous [Mean (Standard Deviation); unit: year] — Age
  year | 52.0 (12.2) | 52.0 (11.2) | 52.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 179 | 345
  Male | 150 | 116 | 266
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 2 | 7
  Black | 108 | 121 | 229
  Latino/Spanish | 6 | 3 | 9
  Other/unknown | 7 | 10 | 17
  White | 190 | 159 | 349
Region of Enrollment [Count of Participants; unit: Participants]
  United States: PA | 247 | 248 | 495
  United States: NJ | 53 | 44 | 97
  United States: Other | 15 | 3 | 18
  United States: Missing | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  College graduate | 172 | 156 | 328
  High school or lower | 34 | 37 | 71
  Some college | 110 | 102 | 212
Employment status [Count of Participants; unit: Participants]
  Homemaker | 15 | 17 | 32
  Student | 3 | 0 | 3
  Employed | 206 | 181 | 387
  Out of work | 36 | 44 | 80
  Retired | 56 | 53 | 109
Annual household income [Count of Participants; unit: Participants]
  > $100,000 | 111 | 77 | 188
  $50,000 - 99,999 | 76 | 95 | 171
  < $50,000 | 103 | 102 | 205
  Missing | 26 | 21 | 47
US residence [Count of Participants; unit: Participants]
  Yes | 315 | 295 | 610
  No | 1 | 0 | 1
Self-rating of health [Count of Participants; unit: Participants]
  Fair | 113 | 110 | 223
  Good | 160 | 133 | 293
  Poor | 17 | 27 | 44
  Very good | 25 | 18 | 43
  Very poor | 1 | 7 | 8
Prior Twitter use [Count of Participants; unit: Participants]
  No | 98 | 101 | 199
  Yes | 218 | 194 | 412
BMI, mean [Mean (Standard Deviation); unit: kg/m^2] | 33.6 (8.5) | 35.0 (10.0) | 34.3 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Activation Measure (PAM) Score From Baseline
Description: The Patient Activation Measure (PAM) is a validated and reliable tool that assesses a person's ability to manage their health, using a 100-point total score scale and four activation levels. The total score ranges from 0 to 100, with higher scores indicating better outcomes-specifically, higher scores represent better outcomes. The overall score is summed from individual items, reflecting the level of activation and self-management ability. The four levels are:
  Level 1 (Score: 0-47.0): Lowest activation, indicating disengagement and lack of confidence in managing health.
  Level 2 (Score: 47.1-55.1): Some awareness of self-management but limited skills and confidence.
  Level 3 (Score: 55.2-67.0): Actively trying to manage health but inconsistent success.
  Level 4 (Score: 67.1-100): Highest activation, indicating confidence and proactive health management.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Twitter Diabetes Control | Twitter Diabetes Intervention
Number analyzed (Participants) | 202 | 129
score on a scale | 3.4 (17.4) | 0.0 (20.7)

2. Secondary Outcome: Change in Systolic Blood Pressure From Baseline
Description: Initial systolic blood pressure (SBP) measurements were obtained from the electronic medical record (EMR). For the majority of patients, final blood pressure measurements (i.e., the 6-month measurement) were obtained in a five to eight month period after enrollment from a documented reading in the the EMR.
  For patients who did not have a documented SBP reading in the health system during this time period, we requested that patients either meet our team in person for a manual reading or provide a photograph from their mobile phone of the screen showing their SBP reading from a home blood pressure cuff, pharmacy machine, or doctor's office from outside of our health system.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Twitter Diabetes Control | Twitter Diabetes Intervention
Number analyzed (Participants) | 252 | 226
mm Hg | -19.8 (19.3) | -18.5 (20.4)

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed
Description: Adverse events were not monitored/assessed
Arm/Group | Twitter Diabetes Control | Twitter Diabetes Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The actual impact of regular tweeting about health may not have been fully actualized in this study. Creating de novo content requires a certain amount of inertia, and prior work shows that individuals engage on social media as passive consumers. The study design was intended to be pragmatic and model real-world use of social media, we did not provide any additional nudges, and although a weekly reminder was useful, participants may have needed feedback on how their tweets were being received.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT02806700/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT02806700/SAP_001.pdf